CLINICAL TRIAL: NCT05523102
Title: Evaluation of Paracetamol as Post-operative Analgetic Modality Compared With Ketorolac
Brief Title: Paracetamol Compared With Ketorolac for Post-operative Analgetic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Radhian Amandito, Pediatrics Resident, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0254
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Pain, Postoperative
Keywords: Acetaminophen; Ketorolac; Postoperative pain; Pediatric; NSAID; Paracetamol; Opioid; Morphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Ketorolac; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Intervention Model Description: Computer generated, randomized selection of patients with 50% probability of assignment into either group Treatment group : paracetamol group Control Group: ketorolac
Who Masked: Participant, Investigator
Masking Description: Patient does not know what analgetics are given, investigator also do not evaluate pain therefore is masked from the intervention given
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Experimental): Paracetamol 15mg/kg 6 hourly for 48 hours post-operatively
  Interventions: Drug: Paracetamol
- Ketorolac (Active Comparator): Ketorolac 0.5mg/kg 8 hourly for 48 hours post-operatively
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Paracetamol — Intravenous paracetamol/acetaminophen
  Other Names: Acetaminophen
  Arms: Paracetamol
Drug: Ketorolac — Intravenous ketorolac/NSAID
  Other Names: NSAID
  Arms: Ketorolac

SUMMARY:
Post-operative analgetic modalities vary between center to center, especially in Indonesia. Considerations include potency/effectivity of the analgetics to achieve adequate pain control as soon as possible, reducing the total opioid dose intake and overall reducing potential opioid adverse effects. NSAID have been known to have more adverse effects than acetaminophen (paracetamol) but offers a higher potency for analgetic effects. Here the investigators compare whether paracetamol is adequate as a post-operative analgetics and confers fewer overall adverse effects when compared with ketorolac (NSAID)

DETAILED DESCRIPTION:
OBJECTIVE: The purpose of this study was to compare the efficacy of Ketorolac versus Paracetamol as an adjunct to Nalbuphine in the management of post-operative pain following elective cardiac surgery.

STUDY DESIGN: Randomized (single-blind) control trial.

SAMPLING TECHNIQUE: Computer generated, randomized selection of patients with 50% probability of assignment into either group.

PLACE AND STUDY DURATION: (single center) PICU and Neurosurgery HCU at the Cipto Mangunkusumo National Referral Center Hospital, Jakarat, Indonesia, over a period of 6 months, from March to August 2022.

METHODS: Eighty-five patients (46 in paracetamol group and 39 in ketorolac group) were randomly assigned to receive either Paracetamol (treatment) or Ketorolac (control), along with the usual pre and intraoperative sedative/analgetics, and opioid as indicated over the first 48 hours postoperatively. The treatment group received injection Paracetamol 15mg/kg six hourly, whereas control group received injection Ketorolac 0.5mg/kg eight hourly.

PRIMARY OUTCOME: The rFLACC (pain score) was evaluated at 0, 8, 12, 24 and 48 hours post-operation and a score of 4 or less was taken as a cut-off for adequate pain control.

SECONDARY OUTCOMES: The total dose of opioid administered to each patient and adverse effects

ELIGIBILITY:
Inclusion Criteria:

* Postoperative patients admitted to Neurosurgery HCU or PICU
* Parents/guardian signed informed consent forms

Exclusion Criteria:

* History of allergy to paracetamol and ketorolac
* Administration of opioid 24 hours before surgery
* Liver dysfunction
* Renal failure

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Pain change | Total 48 hours (0, 8, 12, 24 and 48 hours) post operation
  Post operative analgesic assessment using rFLACC: a pain scoring used primarily for unconscious or disabled children. 0 no pain at all, 10: worst pain (range 0 - 10) Grading is based on the clinical and subjective signs defined in the scoring. For the purposes of this study "adequate pain relief" was defined as achieving a pain score of four or less.

SECONDARY OUTCOMES:
Change in Opioid usage | 48 hours post operatively
  Change in opioid administration as an opioid analgesic
Adverse effects | 48 hours post operatively
  Increase of ALT/AST 3 times above normal range, AKI risk stage, gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Rismala Dewi, Prof, Study Chair — Fakultas Kedokteran Universitas Indonesia; Bernie E Medise, Dr, Study Chair — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No